# A Preliminary Study of Prophylactic Fentanyl Pectin Nasal Spray (FPNS) for Exercise-Induced Breakthrough Dyspnea

Principal investigator: Dr. David Hui

Supportive Care Co-investigators: Dr. Eduardo Bruera, Dr. Suresh Reddy, Dr. Anne

Tsao

Biostatistics Co-investigator: Mr. Gary Chisholm

### **Table of Contents**

| A. Study Objectives | 2 |
|------------------------------------|---|
| B. Background | |
| C. Experimental Approach | |
| D. Statistical Analysis | |
| E. Data Confidentiality Procedures | |
| F. References | |

#### A. Study Objectives

### **Primary objective**

To determine the effect of prophylactic fentanyl pectin nasal spray (FPNS) on the **intensity of exercise-induced breakthrough dyspnea** (numeric rating scale, adjusted for distance walked) between the **first** and **second** 6 minute walk tests. We aim to determine the effect size for both FPNS and placebo arm to inform a larger, adequately powered confirmatory randomized controlled trial.

#### Secondary objectives

- To determine the effect of prophylactic FPNS on the walk distance, neurocognitive function, and adverse effects between the first and second 6 minute walk tests.
- 2. To determine the effect of prophylactic FPNS on the **intensity of dyspnea**, **walk distance**, **neurocognitive function**, **and adverse effects** between the **first** and **third** 6 minute walk tests.
- 3. To compare prophylactic FPNS and placebo on their ability to reduce the intensity of exercise-induced breakthrough dyspnea, walk distance, neurocognitive function, and adverse effects between the first and second 6 minute walk tests, and also between the first and third 6 minute walk tests.

# **B. Background**

**B.1. Significance of Dyspnea.** Dyspnea is a subjective awareness of difficulty breathing, which may be associated with the distressing sensation of suffocation. It is one of the most common and most feared symptoms among cancer patients, occurring in up to 70% of patients in the last 6 weeks of life (Ben-Aharon et al. 2008). Dyspnea is associated with fatigue, anxiety, decreased function and quality of life, and increased mortality (Hauser et al. 2006, Maltoni et al. 2005).

In a study examining 70 patients with dyspnea, 43 (61%) reported breakthrough (episodic or incidental) dyspnea only, 13 (19%) had constant dyspnea only, and 14 (20%) experienced both constant and breakthrough dyspnea. A substantial proportion of the patients with breakthrough dyspnea (18/57, 32%) presented with 5 or more episodes per day, and the majority of episodes lasted <10 minutes (Reddy *et al.* 2009). Breakthrough dyspnea is particularly challenging to treat because of its transient and episodic nature.

Exercise-induced dyspnea (or shortness of breath on exertion) is a subtype of breakthrough dyspnea. This is similar to incident pain (on ambulation) which is a subtype of breakthrough pain. Breakthrough dyspnea has 4 major triggers: exertion, emotional changes, the environment (e.g. altitude, smog), and spontaneous/idiopathic. Because many cancer patients experience severe shortness of breath with activities (i.e. walking), they have to limit their function significantly. In a recent study conducted

by our group, we found that a vast majority of patients (81%) had breakthrough dyspnea. Specifically, dyspnea affects patients' general activity, walking ability, normal work, sleep, mood, relations with others, and enjoyment of life (Reddy *et al.* 2009).

**B.2.** The Current Management of Dyspnea. The current management of dyspnea involves treatment of any reversible causes and supportive measures to minimize the sensation of dyspnea, including treatments such as oxygen, opioids, bronchodilators, and corticosteroids (Ben-Aharon *et al.* 2008, Cranston *et al.* 2008, Jennings *et al.* 2002). A majority of the studies on cancer-related dyspnea so far have focused on patients with dyspnea at rest. In a crossover randomized controlled trial, Bruera *et al.* compared subcutaneous morphine and placebo in 10 patients with advanced cancer who had dyspnea at rest. Subcutaneous morphine was found to be superior to placebo for relief of dyspnea (Bruera *et al.* 1993). This finding was replicated by Mazzocato *et al.* in another randomized controlled trial with similar design (Mazzocato *et al.* 1999). A Cochrane meta-analysis also showed a statistically significant positive effect of opioids on the sensation of breathlessness (p=0.0008), supporting the use of oral or parenteral opioids for treatment of dyspnea in patients with advanced disease (Jennings *et al.* 2002).

Although systemic opioids are established for management of dyspnea at rest, there are currently no evidence-based options for breakthrough dyspnea. In a case series, Bruera et al. reported the use of rescue morphine given subcutaneously for 312 episodes of breakthrough dyspnea in 45 cancer patients. After 30 minutes, 90% reported no to mild dyspnea (Bruera et al. 1993). Based on this study, most clinicians use a dose similar to the rescue opioid dose for breakthrough pain (i.e. 10-20% of total daily dose) to manage breakthrough dyspnea. However, a more recent double-blind randomized controlled trial comparing systemic fentanyl (oral or subcutaneous (SC)), nebulized fentanyl, and nebulized saline for breakthrough dyspnea found no significant difference in dyspnea relief at 10 minutes between the treatment arms (Charles et al. 2008). One of the reasons may be due to the short duration for the primary endpoint (10 minutes). To date, the evidence for opioid use for breakthrough dyspnea remains limited (Table 1). Further research is necessary to improve the management of this distressing and debilitating symptom.

Table 1. Studies of Opioids for Breakthrough Dyspnea

| Study | Methodology and patients | Agent and dose | Outcome |
|---|---|---|---|
| Bruera et al.<br>Ann Intern Med<br>1993 (Bruera et<br>al. 1993) | Prospective case series (45 cancer patients [pts]) | SC morphine 312 doses given (same dose as pain breakthrough) | After 30 minutes, 90% reported no-mild dyspnea; 5% mod-severe dyspnea |
| Benitez-<br>Rosario et al.<br>JPSM 2005<br>(Benitez-<br>Rosario et al.<br>2005) | Retrospective case<br>series (4 cancer<br>pts) | OTFC<br>800mg/1200mcg<br>60mg/800mcg<br>120mg/600mcg<br>15mg/400mcg | RR decreased<br>Dyspnea decreased by 90-<br>100% in 20-60 minutes |

| Sitte et al.<br>JPSM 2008<br>(Sitte and<br>Bausewein<br>2008) | Retrospective case series (1 cancer pt, 2 heart failure pts) | Intranasal fentanyl<br>1/6 of MEDD | RR decreased, improved O <sub>2</sub> saturation in all 3 patients Dyspnea scores not reported |
|---|---|---|---|
| Gauna et al.<br>JPM 2008<br>(Gauna et al.<br>2008) | Prospective case<br>series (2 COPD<br>pts, 2 cancer pts)<br>10 episodes | OTFC<br>30mg/200mcg<br>720mg/400mcg<br>20mg/200mcg<br>24mg/200mcg | RR decreased<br>Dyspnea decreased by 90-<br>100% in 20-60 minutes |
| Charles et al.<br>JPSM 2008<br>(Charles et al.<br>2008) | Prospective,<br>double blind<br>crossover RCT (20<br>cancer pts) | Systemic hydromorphone Nebulized hydromorphone Nebulized saline | Dyspnea decreased similarly in all 3 arms (1.0, 0.9, 0.8) |

Abbreviations: RR=respiratory rate, OTFC=oral transmucosal fentanyl citrate, SC=subcutaneous

B.3. Rapid Onset Opioids for Breakthrough Dyspnea. The episodic and transient nature of breakthrough dyspnea makes fast onset opioids an attractive option. Administration of opioids intravenously or subcutaneously can allow rapid delivery of the drug, although many patients do not have access to these routes at home. Fentanyl is a highly lipophilic compound. Over the past decade, there has been active development of fentanyl, including delivery by the transmucosal (oral transmucosal fentanyl citrate [OTFC], Actig), buccal (Fentora) and intranasal (Lazanda, Instanyl) formulations (Gordon and Schroeder 2008, Lecybyl and Hanna 2007). These fentanyl formulations have been successfully used to manage breakthrough pain (Christie et al. 1998, Coluzzi et al. 2001, Fallon et al. 2011, Farrar et al. 1998, Mercadante et al. 2007, Portenov et al. 1999, Portenoy et al. 2006, Portenoy et al. 2010, Slatkin et al. 2007), although their role in breakthrough dyspnea has only been reported in a handful of studies. Two small retrospective case series reported on the use of transmucosal and intranasal fentanyl (Benitez-Rosario et al. 2005, Sitte and Bausewein 2008) and one prospective series examined the use of OTFC (Gauna et al. 2008) suggest significant improvement in breakthrough dyspnea with these agents. Randomized controlled trials are urgently needed to confirm these findings with rapid onset opioids, which could potentially open up a new therapeutic indication for these medications.

FPNS is a particularly attractive option for breakthrough dyspnea. It was approved by the US Food and Drugs Administration (FDA) in 2011 for breakthrough pain in opioid-tolerant patients with cancer, and represents an alternative delivery system for fentanyl in addition to the transdermal, parenteral, and transmucosal routes. Pharmacokinetic studies revealed that FPNS has a bioavailability of approximately 80% (Fisher et al. 2010, Fisher et al. 2010). The time to maximal effect (Tmax) was between 15-20 minutes (Fisher et al. 2010, Fisher et al. 2010). FPNS has been found in clinical trials to provide greater and more rapid pain relief and reduces pain better than placebo (Kress et al. 2009) and transmucosal fentanyl citrate (Mercadante et al. 2009).

# C. Experimental Approach

C.1. Overall Study design. This is an investigator initiated study supported in part by Depomed, Inc. We propose a 2arm, double blind, parallel randomized controlled trial of FPNS and placebo for cancer patients with breakthrough dyspnea (Figure 1). The main goal of this study is to determine the effect size for both FPNS and placebo arm to inform a larger, adequately powered confirmatory randomized controlled trial. After study consent, eligible patients will be asked to complete a number of surveys and a 6minute walk test at baseline, rest until they return to baseline dyspnea, and then do a second 6-minute walk test 20 minutes after they have been given either FPNS or placebo prophylactically. They will then rest again to return to baseline dyspnea, and then do another 6-minute walk test 20 minutes after repeating the same dose of either FPNS or placebo (with at least 30 minutes between the first



Figure 1. Study Flow Chart

and second dose). This design will allow testing of both single and repeated dosing on dyspnea under a double blind design.

Based on our experience conducting symptom control trials, this study will take between 1.5-2 hours to complete on a single visit. We believe this study design is feasible and would not add undue burden for patients. Patients will be compensated with a \$50 gift card for their time and effort.

**C.2. Eligibility Criteria.** The eligibility criteria are shown in Table 2. **Table 2. Study Eligibility Criteria** 

#### **Inclusion Criteria**

- 1. Diagnosis of cancer
- 2. Breakthrough dyspnea, defined in this study as dyspnea on exertion with an average intensity level >=3/10 on the numeric rating scale
- Outpatient at MD Anderson Cancer Center seen by the Supportive Care Service or Thoracic Medical Oncology
- 4. Ambulatory and able to walk with or without walking aid
- 5. On strong opioids with morphine equivalent daily dose of 80-500 mg, with stable (i.e. +/- 30%) regular dose over the last 24 hours
- 6. Karnofsky performance status >=50%
- 7. Age 18 or older
- 8. Able to complete study assessments

#### **Exclusion Criteria**

- 1. Dyspnea at rest >=7/10 at the time of enrollment
- 2. Supplemental oxygen requirement >6 L per minute
- 3. Delirium (i.e. Memorial delirium rating scale >13)
- 4. History of unstable angina or myocardial infarction 1 month prior to study enrollment
- 5. Resting heart rate >120 at the time of study enrollment
- 6. Systolic pressure >180 mmHg or diastolic pressure >100 mmHg at the time of study enrollment
- 7. History of active opioid abuse within the past 12 months
- 8. History of allergy to fentanyl
- 9. Unwilling to provide informed consent
- 10. Patients who currently have no evidence of disease
- **C.3. Study screening.** A 2 step consent process will be used. First, a verbal consent will be obtained by the study staff to proceed with screening of potential participants for eligibility and to characterize their dyspnea using the dyspnea survey and the cancer dyspnea scale. Outpatients may be contacted by phone within 1 week prior to their scheduled clinic visit to informed them of this study so they can make necessary arrangements if interested in participating. Eligible patients will then be formally enrolled onto the study after they have signed the informed consent indicating a willingness for the patient to participate in the trial. The number of patients screened, approached, eligible and enrolled will be documented. Reasons for refusal for eligible patients will also be captured. Based on our experience with similar trials, we expect that a majority of patients will complete this study.
- **C.4. Randomization.** A computer generated sequence in permuted blocks will be used to assign patients to either FPNS or placebo and provided via a secured website, stratified by baseline level of dyspnea NRS at rest at the time of enrollment (i.e. 0-3, 4-6). Biostatistics will set up a Randomization website. Investigational Pharmacy personnel will perform the randomization assignment.
- **C.5. Blinding.** Both patients and the research staff conducting the assessment will be blinded to the treatment assignment. FPNS will be dispensed by Dispensing Pharmacy at MD Anderson. Placebo will be identical in appearance to the FPNS.
- **C.6. Research staff.** An orientation will be held with research staff involved in this study to introduce them with the study design, and standardize the provision of each intervention.
- **C.7. Study Interventions.** The supply of study medication (both FPNS and placebo) will be provided by Depomed, Inc. FPNS is FDA approved (NDA 022569/S-007) for treatment of breakthrough cancer pain in opioid-tolerant patients. Immediately upon patient enrollment, the study physician will be notified and will determine the morphine equivalent daily dose (MEDD) in real time using standardized equianalgesic ratios.

Based on clinical practice and similarly to the dose used for breakthrough pain, we will use an FPNS dose equivalent to 15-25% of the MEDD (Table 3). For patients randomized to receive FPNS, the study medication will be provided by Dispensing Pharmacy and will then be administered intranasally 20 minutes before the second 6-minute walk test. The same dose will be repeated at least 30 minutes after the first dose and 20 minutes prior to the third and final 6 minute walk test. We estimated the FPNS dose based on the following assumptions:

- A rescue dose of 15-25% of the MEDD is safe and adequate for relief of dyspnea (Bruera *et al.* 1993, Charles *et al.* 2008).
- FPNS has approximately 80% oral bioavailability (Fisher et al. 2010, Fisher et al. 2010).
- With repeat dosing 30 minutes apart, the maximum concentration (Cmax) for FPNS is approximately 1.6x higher than the first dose.

The modeled pharmacokinetic data for repeated dosing 30 minutes apart is shown in Figure 2. As a precautionary measure, patients will be asked to wait for 1 hour after completing the last walk before leaving MD Anderson. At the end of 1 hour, they will be assessed by our research staff before being released. If excessive drowsiness or adverse events occur, the study physician will assess the patients.



Figure 2. Modeled Pharmacokinetic Data on Repeat Dosing of Fentanyl Pectin Nasal Spray after 30 m

Table 3. Dose of Fentanyl Pectin Nasal Spray Based on Morphine Equivalent Daily Dose<sup>a</sup>

| Morphine | Total Fentanyl | Number of | Number of |
|------------------|------------------|-------------|----------------|
| equivalent daily | Pectin Nasal | FPNS sprays | Placebo sprays |
| dose (mg) | Spray Dose (mcg) | | |

| | | | | Page 8 of 13 |
|---|---|---|---|---|
| 80-159 | 100 | 1 (100 mcg in one nostril) | 1 | |
| 160-239 | 200 | 2 (100 mcg in each nostril) | 2 | |
| 240-319 | 300 | 3 (100 mcg in one nostril<br>and 2 x 100 mcg in the<br>other nostril) <sup>b</sup> | 3 | |
| 320-540 | 400 | 4 (2 x 100 mcg in each nostril) | 4 | |

<sup>&</sup>lt;sup>a</sup> FPNS is available in 100 mcg.

Placebo will be identical in appearance to the FPNS, and given to patients 20 minutes before the second and the third 6-minute walk test. Both the patient and the research staff conducting the assessments will be blinded to the nature of the intervention. During this entire study, patients will be monitored closely by trained research staff, and will have rapid access to medical care if needed.

Because this involves only 2 doses given to opioid tolerant patients, and under close monitoring by trained staff, we believe the dosing schedule proposed is safe.

- **C.8. Medication use during study.** To minimize the co-intervention effect on dyspnea, patients will be advised to avoid using breakthrough opioids (for any reason) or bronchodilators for at least 2 hours prior to and during the study.
- **C.9. The 6-minute walk tests** will be conducted based on guidelines from the American Thoracic Society (Laboratories 2002). Walking aid and supplemental oxygen via nasal prongs are allowed as long as patients keep them the same as before enrollment and during the entire study. This walking test allows patients to rest if they need to, and is highly acceptable to patients. It provides important information regarding patients' functional status, exercise capacity, and health-related quality of life (Guyatt *et al.* 1985, Guyatt *et al.* 1985). Before and after each test, we will be assessing the (1) dyspnea level with numeric rating scale and Borg scale, and the (2) respiratory rate and oxygen saturation. After each test, we will also be assessing (1) the distance walked at the end of each minute or portion of, (2) the total walking time, (3) the level of dyspnea at the end of each minute or portion of (NRS and Borg scale), and (4) the average walking speed.

The 6-minute walk test has excellent short term reproducibility (Guyatt *et al.* 1985), as well as good face, construct, and predictive validity (Du Bois *et al.* 2011), and changes in this test are concordant with changes in symptoms and mortality (Olsson *et al.* 2005). The minimal clinical significant difference is found to be 24-45 m for patients with idiopathic pulmonary fibrosis (Du Bois *et al.* 2011), and 86 m for patients with COPD.

The first 6-minute walk test was designed to provide important information regarding a patient's level of dyspnea on exertion, and to facilitate intra-individual comparison since there is significant variability in the expression of dyspnea among patients.

<sup>&</sup>lt;sup>b</sup> For the 300 mcg dose, patients will receive 1 spray in each nostril, then another spray again in the one of the nostrils.

- **C.10. Variable rest period.** After the first and second 6 minute walk test, patients will be asked to sit down and rest. How long they rest would depend on when they return to baseline level of dyspnea numeric rating score + 1 or below (e.g. if baseline dyspnea = 4, they need to return to a level of 5 or less to qualify for next stage). During this rest period, patients will be assessed every 5 minutes to check their dyspnea level. If their dyspnea level met criteria and they feel ready to walk again, they will be given the study treatment and asked to wait for 20 minutes before they walk. At least 30 minutes should elapse between each dose of the study medication.
- **C.11. Stopping rules.** Patients who do not develop any increase from their baseline dyspnea after the first 6-minute walk will not proceed to the next stage because of the lack of exercise induced dyspnea. If at any time during the study patients develop chest pain, severe leg cramps, staggering, diaphoresis, and/or dizziness, they will be asked to stop the study. If patients require more than 1 hour of rest and their dyspnea level still has not returned to baseline, they will also be taken off study. We plan to replace these patients and any other individuals who are not evaluable because they have not started the 2nd walk test.

**C.12. Study assessments.** See Table 4 for a detailed description of all study assessments.

**Table 4. Summary of Study Assessments** 

| Assessments | Base-<br>line | Post<br>1 <sup>st</sup><br>6MWT | Rest<br>#1 | Pre<br>2 <sup>nd</sup><br>6MW | Post<br>2 <sup>nd</sup><br>6MW | Rest<br>#2 | Pre<br>3 <sup>rd</sup><br>6MW | Post<br>3 <sup>rd</sup><br>6MW |
|---|---|---|---|---|---|---|---|---|
| Demographics and cancer | ✓ | | | | | | | |
| diagnosis <sup>1</sup> | | | | | | | | |
| Medication history <sup>2</sup> | $\checkmark$ | | | | | | | |
| Karnofsky performance status <sup>3</sup> | $\checkmark$ | | | | | | | |
| Edmonton Symptom Assessment | $\checkmark$ | | | | | | | |
| Scale <sup>4</sup> | | | | | | | | |
| Dyspnea Survey <sup>5</sup> | $\checkmark$ | | | | | | | |
| Cancer Dyspnea Scale <sup>6</sup> | $\checkmark$ | | | | | | | |
| O <sub>2</sub> saturation and respiratory rate | $\checkmark$ | $\checkmark$ | | $\checkmark$ | $\checkmark$ | | $\checkmark$ | $\checkmark$ |
| Dyspnea Numeric Rating Scale <sup>7</sup> | $\checkmark$ | $\checkmark$ | $\checkmark$ | $\checkmark$ | $\checkmark$ | $\checkmark$ | $\checkmark$ | $\checkmark$ |
| Dyspnea Borg scale <sup>8</sup> | $\checkmark$ | $\checkmark$ | $\checkmark$ | $\checkmark$ | $\checkmark$ | $\checkmark$ | $\checkmark$ | $\checkmark$ |
| Walking test parameters9 | | $\checkmark$ | | | $\checkmark$ | | | ✓ |
| Adverse effects <sup>10</sup> | | | | $\checkmark$ | $\checkmark$ | | $\checkmark$ | $\checkmark$ |
| Neurocognitive testing <sup>11</sup> | | $\checkmark$ | | | $\checkmark$ | | | ✓ |
| Global assessment <sup>12</sup> | | | | | $\checkmark$ | | | $\checkmark$ |
| Blinding <sup>13</sup> | | | | | | | | $\checkmark$ |
| Patient satisfaction <sup>14</sup> | | | | | | | | $\checkmark$ |

<sup>&</sup>lt;sup>1</sup> patient initials, medical record number, date of birth, sex, race, education, marital status, cancer diagnosis, co-morbidities, cause(s) of dyspnea.

<sup>&</sup>lt;sup>2</sup> medications that could be used to treat dyspnea, including scheduled and as needed opioids, bronchodilators, and steroids will be documented.

<sup>&</sup>lt;sup>3</sup> an 11-point assessment scale that rates patients' functional status between 0% (death) and 100% (completely asymptomatic) based on their ambulation, activity level, and disease severity (Schag *et al.* 1984).

<sup>&</sup>lt;sup>4</sup> validated questionnaire that measures 10 common symptoms in the past 4 hours (pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, appetite, sleep, and feeling of well being) using numeric rating scales (Bruera *et al.* 1991).

- <sup>5</sup> characterization of patients dyspnea including the following: presence of dyspnea at rest, average dyspnea in last 24 hours, worse dyspnea in last 24 hours, best dyspnea in last 24 hours, number of episodes of exacerbation per day, triggers of breakthrough dyspnea, average duration of each episode, current treatment for breakthrough dyspnea.
- <sup>6</sup> validated 12-item questionnaire specifically designed to assess the quality of dyspnea in cancer patients during the past few days (Tanaka *et al.* 2000). Each item has a score between 1 and 5, for a maximum of 60. There are sub-scores for sense of effort, anxiety, and discomfort.
- <sup>7</sup> a 0 (no dyspnea) to 10 (worst dyspnea) categorical scale validated for rating the severity of dyspnea (Dorman *et al.* 2007, Gift and Narsavage 1998, Powers and Bennett 1999). We will be measuring it every minute during the 6 minute walk test at 0, 1 min, 2 min, 3 min, 4 min, 5 min and 6 min (or end of walk).
- <sup>8</sup> a 0 to 10 categorical scale for rating the severity of dyspnea. It is a ratio scale with descriptive anchors throughout the range in which a rating of 8 signifies breathlessness twice as severe as 4, which in turn is twice as severe as 2 (Dorman *et al.* 2007, Gift and Narsavage 1998, Kendrick *et al.* 2000, Powers and Bennett 1999). We will be measuring it 0 and 6 min (or end of walk) of each walk. The NRS will be administered before modified Borg scale.
- <sup>9</sup> include the total distance walked, total walking time, the distance and time of first rest due to dyspnea, average walking speed.
- <sup>10</sup> adverse effects related to the use of FPNS, such as dizziness, drowsiness, nausea, stuffy/blocked nose, runny nose, itching/sneezing, nose dryness, cough, sore throat, and taste disturbance will be assessed using a numeric rating scale from 0-10.
- <sup>11</sup> patients will be asked to do finger tapping 10 and 30 sec, arithmetic, reverse memory of digits, and visual memory). This has been used in other studies by our group (Bruera *et al.* 1992) <sup>12</sup> patients will be asked about their dyspnea (worse, about the same, or better) comparing between the level of dyspnea between the first and second 6-minute walk tests (Guyatt *et al.* 1993, Redelmeier *et al.* 1996).
- <sup>13</sup> blinding will be done by asking patients which group assignment they received: "FPNS", "placebo", or "do not know".
- <sup>14</sup> study satisfaction is assessed with the following questions, "Was it worthwhile for you to participate in this research study?", "If you had to do it over, would you participate in this research study again?", "Would you recommend participating in this research study to others?", "Did you quality of life get better by participating in this research study?", "Did you quality of life get worse by participating in this research study?"
- **C.13. Feasibility data.** In addition to clinical outcomes, we will also collect feasibility data in this study Rates of recruitment and retention (% of subjects able to complete the study)
- Reasons for refusal and dropout
- Outcome measure—we will compare the sensitivity of Numeric rating scale and Borg scale to change, and identify key measure for future study
- Participant satisfaction—participants will provide an opinion regarding their satisfaction with study overall
- **C.14.** Patient Safety, Monitoring, and Confidentiality. During the study, trained research staff will be performing study assessments and monitoring the patients carefully throughout the study period. A study physician will also be available by pager to address any concerns, distress or questions, and will attend to the patient as needed. Patients will be doing the test in a hallway outside the Supportive Care Center which typically does not have a lot of traffic, and will have immediate access to medical and nursing care if needed. See stopping rules below for further details. With the planned

doses of fentanyl in opioid-tolerant patients, we do not expect any significant side effects.

Regulatory monitoring will be provided by the principal investigator, the Institutional Review Board (IRB), and the Data Safety and Monitoring Board (DSMB). Patient confidentiality will be ensured by use of study numbers, secure storage of clinical data, and anonymous reporting.

#### **D. Statistical Analysis**

- **D.1. Sample Size Calculation.** Patients who have started the second walk test will be considered evaluable for this study's primary endpoint. 10 evaluable patients in the fentanyl arm provides 80% power to detect an effect size as small as 1.0 when alpha=5% using a two-sided paired t-test to compare dyspnea between the first and second walk tests. Results from this study will be used to calculate the sample size for an adequately powered randomized controlled trial.
- **D.2. Data Analysis.** Summary descriptive statistics will be provided for demographics, outcomes, and other collected variables and will include proportions, medians, means, 95% confidence intervals, and other simple statistics as appropriate for the measure. Comparisons within arms will be performed using paired t-tests or signed rank tests.

#### **E. Data Confidentiality Procedures**

Health information will be protected and we will maintain the confidentiality of the data obtained from the patient's chart.

Collection of identifiers: We will collect and securely store patients' identifiers (including name, medical record number and demographic specifications). Each patient will be assigned a study number that will be the only identifier to figure in the analytical file and personal data will not be disclosed in any form. The key linking these numbers will be retained in a securely locked file by the investigator.

Data Storage: Protection of electronic and paper records will be guaranteed. All electronic records will be stored on password-protected institution computers behind the institution firewall. Any paper records will be classified and stored in locked files inside a locked office.

Training of personnel: Only MDACC personnel trained in maintaining confidentiality, the principle investigators and co-investigators, will have access to study records.

Data sharing: Study data will not be shared with any individuals or entities. The data will be kept by the principle investigator in a locked file cabinet.

Final disposition of study records: These data will be used only for this research study data files will be destroyed 5 years after publication of the findings.

#### F. References

- 1. Ben-Aharon I, Gafter-Gvili A, Paul M, et al. Interventions for alleviating cancer-related dyspnea: A systematic review. *J Clin Oncol* 2008;26:2396-404.
- 2. Benitez-Rosario MA, Martin AS, Feria M. Oral transmucosal fentanyl citrate in the management of dyspnea crises in cancer patients. *J Pain Symptom Manage* 2005;30:395-7.
- 3. Bruera E, Kuehn N, Miller MJ, et al. The edmonton symptom assessment system (esas): A simple method for the assessment of palliative care patients. *J Palliat Care* 1991;7:6-9.

- 4. Bruera E, Miller MJ, Macmillan K, et al. Neuropsychological effects of methylphenidate in patients receiving a continuous infusion of narcotics for cancer pain. *Pain* 1992;48:163-6.
- 5. Bruera E, MacEachern T, Ripamonti C, et al. Subcutaneous morphine for dyspnea in cancer patients. *Ann Intern Med* 1993;119:906-7.
- 6. Charles MA, Reymond L, Israel F. Relief of incident dyspnea in palliative cancer patients: A pilot, randomized, controlled trial comparing nebulized hydromorphone, systemic hydromorphone, and nebulized saline. *J Pain Symptom Manage* 2008;36:29-38.
- 7. Christie JM, Simmonds M, Patt R, et al. Dose-titration, multicenter study of oral transmucosal fentanyl citrate for the treatment of breakthrough pain in cancer patients using transdermal fentanyl for persistent pain. *J Clin Oncol* 1998;16:3238-45.
- 8. Coluzzi PH, Schwartzberg L, Conroy JD, et al. Breakthrough cancer pain: A randomized trial comparing oral transmucosal fentanyl citrate (otfc) and morphine sulfate immediate release (msir). *Pain* 2001;91:123-30.
- 9. Cranston JM, Crockett A, Currow D. Oxygen therapy for dyspnoea in adults. *Cochrane Database Syst Rev* 2008.
- 10. Dorman S, Byrne A, Edwards A. Which measurement scales should we use to measure breathlessness in palliative care? A systematic review. *Palliat Med* 2007;21:177-91.
- 11. du Bois RM, Weycker D, Albera C, et al. Six-minute-walk test in idiopathic pulmonary fibrosis: Test validation and minimal clinically important difference. *Am J Respir Crit Care Med* 2011;183:1231-7.
- 12. Fallon M, Reale C, Davies A, et al. Efficacy and safety of fentanyl pectin nasal spray compared with immediate-release morphine sulfate tablets in the treatment of breakthrough cancer pain: A multicenter, randomized, controlled, double-blind, double-dummy multiple-crossover study. *J Support Oncol* 2011;9:224-31.
- 13. Farrar JT, Cleary J, Rauck R, et al. Oral transmucosal fentanyl citrate: Randomized, double-blinded, placebo-controlled trial for treatment of breakthrough pain in cancer patients. *J Natl Cancer Inst* 1998;90:611-6.
- 14. Fisher A, Watling M, Smith A, et al. Pharmacokinetic comparisons of three nasal fentanyl formulations; pectin, chitosan and chitosan-poloxamer 188. *Int J Clin Pharmacol Ther* 2010;48:138-45.
- 15. Fisher A, Watling M, Smith A, et al. Pharmacokinetics and relative bioavailability of fentanyl pectin nasal spray 100 800 microg in healthy volunteers. *Int J Clin Pharmacol Ther* 2010;48:860-7.
- 16. Gauna AA, Kang SK, Triano ML, et al. Oral transmucosal fentanyl citrate for dyspnea in terminally ill patients: An observational case series. *J Palliat Med* 2008;11:643-8.
- 17. Gift AG, Narsavage G. Validity of the numeric rating scale as a measure of dyspnea. *Am J Crit Care* 1998;7:200-4.
- 18. Gordon D, Schroeder M. Oral transmucosal fentanyl citrate--otfc (actiq) #103. *J Palliat Med* 2008;11:633-4.
- 19. Guyatt GH, Sullivan MJ, Thompson PJ, et al. The 6-minute walk: A new measure of exercise capacity in patients with chronic heart failure. *Can Med Assoc J* 1985;132:919-23.
- 20. Guyatt GH, Thompson PJ, Berman LB, et al. How should we measure function in patients with chronic heart and lung disease? *J Chronic Dis* 1985;38:517-24.
- 21. Guyatt GH, Feeny DH, Patrick DL. Measuring health-related quality of life. *Ann Intern Med* 1993:118:622-9.
- 22. Hauser CA, Stockler MR, Tattersall MH. Prognostic factors in patients with recently diagnosed incurable cancer: A systematic review. *Support Care Cancer* 2006;14:999-1011.
- 23. Jennings AL, Davies AN, Higgins JP, et al. A systematic review of the use of opioids in the management of dyspnoea. *Thorax* 2002;57:939-44.

- 24. Kendrick KR, Baxi SC, Smith RM. Usefulness of the modified 0-10 borg scale in assessing the degree of dyspnea in patients with copd and asthma. *Journal of emergency nursing: JEN:* official publication of the Emergency Department Nurses Association 2000;26:216-22.
- 25. Kress HG, Oronska A, Kaczmarek Z, et al. Efficacy and tolerability of intranasal fentanyl spray 50 to 200 microg for breakthrough pain in patients with cancer: A phase iii, multinational, randomized, double-blind, placebo-controlled, crossover trial with a 10-month, open-label extension treatment period. *Clin Ther* 2009;31:1177-91.
- 26. Laboratories ATSCoPSfCPF. Ats statement: Guidelines for the six-minute walk test. *Am J Respir Crit Care Med* 2002;166:111-7.
- 27. Lecybyl R, Hanna M. Fentanyl buccal tablet: Faster rescue analgesia for breakthrough pain? *Future oncology (London, England)* 2007;3:375-9.
- 28. Maltoni M, Caraceni A, Brunelli C, et al. Prognostic factors in advanced cancer patients: Evidence-based clinical recommendations--a study by the steering committee of the european association for palliative care. *J Clin Oncol* 2005;23:6240-8.
- 29. Mazzocato C, Buclin T, Rapin CH. The effects of morphine on dyspnea and ventilatory function in elderly patients with advanced cancer: A randomized double-blind controlled trial. *Ann Oncol* 1999;10:1511-4.
- 30. Mercadante S, Villari P, Ferrera P, et al. Transmucosal fentanyl vs intravenous morphine in doses proportional to basal opioid regimen for episodic-breakthrough pain. *Br J Cancer* 2007;96:1828-33.
- 31. Mercadante S, Radbruch L, Davies A, et al. A comparison of intranasal fentanyl spray with oral transmucosal fentanyl citrate for the treatment of breakthrough cancer pain: An open-label, randomised, crossover trial. *Curr Med Res Opin* 2009;25:2805-15.
- 32. Olsson LG, Swedberg K, Clark AL, et al. Six minute corridor walk test as an outcome measure for the assessment of treatment in randomized, blinded intervention trials of chronic heart failure: A systematic review. *Eur Heart J* 2005;26:778-93.
- 33. Portenoy RK, Payne R, Coluzzi P, et al. Oral transmucosal fentanyl citrate (otfc) for the treatment of breakthrough pain in cancer patients: A controlled dose titration study. *Pain* 1999:79:303-12.
- 34. Portenoy RK, Taylor D, Messina J, et al. A randomized, placebo-controlled study of fentanyl buccal tablet for breakthrough pain in opioid-treated patients with cancer. *The Clinical Journal of Pain* 2006;22:805-11.
- 35. Portenoy RK, Raffaeli W, Torres LM, et al. Long-term safety, tolerability, and consistency of effect of fentanyl pectin nasal spray for breakthrough cancer pain in opioid-tolerant patients. *J Opioid Manag* 2010;6:319-28.
- 36. Powers J, Bennett SJ. Measurement of dyspnea in patients treated with mechanical ventilation. *Am J Crit Care* 1999;8:254-61.
- 37. Reddy SK, Parsons HA, Elsayem A, et al. Characteristics and correlates of dyspnea in patients with advanced cancer. *J Palliat Med* 2009;12:29-36.
- 38. Redelmeier DA, Guyatt GH, Goldstein RS. Assessing the minimal important difference in symptoms: A comparison of two techniques. *J Clin Epidemiol* 1996;49:1215-9.
- 39. Schag CC, Heinrich RL, Ganz PA. Karnofsky performance status revisited: Reliability, validity, and guidelines. *J Clin Oncol* 1984;2:187-93.
- 40. Sitte T, Bausewein C. Intranasal fentanyl for episodic breathlessness. *J Pain Symptom Manage* 2008;36:e3-6.
- 41. Slatkin NE, Xie F, Messina J, et al. Fentanyl buccal tablet for relief of breakthrough pain in opioid-tolerant patients with cancer-related chronic pain. *J Support Oncol* 2007;5:327-34.
- 42. Tanaka K, Akechi T, Okuyama T, et al. Development and validation of the cancer dyspnoea scale: A multidimensional, brief, self-rating scale. *Br J Cancer* 2000;82:800-5.